CLINICAL TRIAL: NCT00646867
Title: An Open Label Study of the Therapeutic Effects of Tetrix Cream in Allergic Contact and Irritant Contact Dermatitis
Brief Title: Effect of Tetrix on Alleviation of Burning,Itching Associated With Lesions of Contact Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coria Laboratories, Ltd. (Industry)
Responsible Party: D. Innes Cargill, PhD, Coria Laboratories, Ltd.
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 805 806 09 004
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Contact Dermatitis
Keywords: Tetrix cream, contact dermatitis, effect on burning and itching
MeSH Terms: conditions — Dermatitis, Contact; Pruritus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Experimental
  Interventions: Device: Tetrix
- 2 (Placebo Comparator): Placebo
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Tetrix — Twice daily topical application
  Arms: 1
Device: Placebo — Twice daily topical application
  Arms: 2

SUMMARY:
To determine if Tetrix Cream, when applied to the skin lesions on patients with contact dermatitis, improves the symptoms of burning and itching.

ELIGIBILITY:
Inclusion Criteria:

1. Normal subjects with sensitivity to nickel
2. Subjects with hand eczema

Exclusion Criteria:

under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Improvement in symptoms of burning and itching. | after 14 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Fowler, MD, Principal Investigator — Dermatology Specialists, LLC
Locations (1):
- Dermatology Specialists, LLC, Louisville, Kentucky, United States